CLINICAL TRIAL: NCT02377271
Title: Effect of Bosentan in Patients With Non Arteritic Ischemic Optic Neuropathy
Brief Title: ENDOTHELION Study Group: Effect of Bosentan in NAION Patients
Acronym: ENDOTHELION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-000848-14
Record Dates: First submitted 2014-12-05; First posted 2015-03-03 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-04

CONDITIONS: Ischemic Optic Neuropathy
Keywords: Bosentan
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bosentan (Experimental): Bosentan at a dose of 125 mg two times daily, will be administered orally, twice a day, during eight weeks
  Interventions: Drug: bosentan
- Placebo (Placebo Comparator): placebo drug , twice a day, during eight weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bosentan — treatment by bosentan or placebo is randomized , 125 mg twice a day
  Arms: Bosentan
Drug: placebo — treatment by bosentan or placebo is randomized
  Arms: Placebo

SUMMARY:
Acute ischemic optic neuropathy are the second leading cause of optic neuropathy after glaucoma in the population aged over 50 years. The visual prognosis of the condition is unfavorable in the great majority of cases, with significant effects on the visual field and vision. The severity of the unilateral condition is also associated with bilateralization in 15% at 5 years. There is no effective treatment for the acute phase of the disease or to reduce the rate of bilateralization. In this context, it is essential to develop new therapeutic strategies in the acute phase of the disease to reduce the anatomical optic nerve damage.

DETAILED DESCRIPTION:
The main objective of our study will be to compare the treatment with bosentan to placebo for 8 weeks for recovery anatomical criteria (RFNL in OCT, optic atrophy) and functional (visual acuity, visual field). The primary endpoint will be the improvement of the visual field, a major criterion of the affected visual function in this disease.

The evaluation of bosentan will mainly after 8 weeks of treatment in order to assess the effectiveness of drug treatment in the absence of continuous positive airway pressure (set up after three months if necessary, feasible confounding factor for the evaluation of results ), the period of three months is sufficient to assess the anatomical and functional recovery (disappearance of papilledema).

ELIGIBILITY:
Inclusion Criteria:

* Non arteritic ischemic optic neuropathy (NAION) with onset < 21 days
* Age ≥ 50 years old
* Signed informed consent form
* Patients affiliated with a national health insurance scheme or beneficiaries of such a scheme

Exclusion Criteria:

* Pregnant women, women in labour or breast-feeding mother
* Patients with other acute or chronic intercurrent ocular pathology interfering with visual acuity or visual field (diabetes, drug-induced or other retinopathy, other optic neuropathy including uni- or contralateral glaucoma and/or intraocular pressure > 30 mmHg, advanced cataract, corneal opacities, amblyopia < 5/10, severe myopia > -6 diopters, retinal disease)
* Simultaneous bilateral NAAION, 1 month apart or less
* Signs that may raise suspicion of other inflammatory neuropathy: arterial NAAION (Horton's disease), pain on eye movement or any signs suggestive of optic neuritis, known diagnosis of multiple sclerosis, history of inflammatory optic neuropathy (homo- or ipsi-lateral). A temporal artery biopsy should be performed if there are symptoms suggestive of Horton's disease, or if there is pale and/or diffuse edema, or obliteration of the associated central retinal artery.
* Patients with systolic blood pressure below 100 mmHg
* Patient with orthostatic hypotension (20 mmHg drop in SBP and/or 10 mmHg drop in DBP when moving to a standing position)
* Neurological history of vascular or tumour-related changes to the visual field or other optic neuropathy
* Systemic inflammatory disease
* Known allergy to bosentan
* Patients with moderate to severe hepatic impairment (Child-Pugh class B or C), biliary cirrhosis (serum levels of liver aminotransferases, aspartate aminotransferases (ASAT) and/or alanine aminotransferases (ALAT), greater than three times the upper limit of normal, bilirubin greater than twice normal)
* Estimated glomerular filtration rate (GFR) < 30 ml/min/1.73 m2
* Patients treated with drugs whose efficacy may be reduced by activation of cytochrome P450, 2C9, 3A4 and 2C19 isoenzymes
* Patients treated with amiodarone
* Patient treated with systemic corticosteroids (background treatment or treatment initiated at the time of NAAION diagnosis)
* Person deprived of liberty by judicial or administrative decision, adult protected by law, hospitalized person
* Ongoing participation in another clinical research study or in the exclusion period of another clinical study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
mean deviation of automated visual field | 3 month
  Humphrey 30-2 SITA-standard

SECONDARY OUTCOMES:
visual acuity | 6, 12 and 24 month
  ETDRS scale
optic nerve fiber layer thickness | 3, 6, 12 and 24 month
  OCT measurement
mean deviation of automated visual field for healthy eye and NAION eye | 3, 6, 12 and 24 month
  Humphrey 30-2
inflammatory marker and prepro-endothelin dosing | 3 month
  RANTES, MCP-1, TNF-α, INF-γ, IL-6, IL-10 and TGF-β
mean deviation of automated visual field for controlateral eye | 24 month
  Humphrey 30-2 sita-standard
VFQ-25 score | 3 and 12 month
  VFQ-25 quality of life
rate of bilateral occurence of NAION | at 24 month visit
  rate of bilateralization

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Pr CHIQUET, Prof, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (7):
- France (7):
  - University Hospital of Angers, Angers
  - University Hospital of Bordeaux, Bordeaux
  - CHU de Grenoble, Grenoble
  - University Hospital of Grenoble Michallon, Grenoble
  - Ophtalmological fondation of Rothschild + Bichat Hospital, Paris
  - Centre National d'Ophtalmologie XV-XX, Paris
  - University hospital of Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiquet C, Vignal C, Gohier P, Heron E, Thuret G, Rougier MB, Lehmann A, Flet L, Quesada JL, Roustit M, Milea D, Pepin JL; ENDOTHELION group. Treatment of nonarteritic anterior ischemic optic neuropathy with an endothelin antagonist: ENDOTHELION (ENDOTHELin antagonist receptor in Ischemic Optic Neuropathy)-a multicentre randomised controlled trial protocol. Trials. 2022 Oct 29;23(1):916. doi: 10.1186/s13063-022-06786-9. PMID 36309759